CLINICAL TRIAL: NCT04507815
Title: Combined tDCS and Cognitive Training for Mild Cognitive Impairment (MCI) and Early Clinical Alzheimer's Type Dementia (CATD)
Brief Title: tDCS and Cognitive Training for Mild Cognitive Impairment and Alzheimer's Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Casey Gilmore, PhD, Research Scientist, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAM-20-00623
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): Participants will receive 10 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over left frontal cortex, cathode over right frontal cortex; 2 mAmps for 20 minutes).
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Participants will receive 10 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 secs, then immediately ramped back down. This ramp up/down method is done at the end of the stimulation period, as well. This method mimics the physical sensation of stimulation typically encountered at the very beginning and end of the intervention period.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the left frontal cortex for 20 minutes.
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning and end of session).
  Arms: Sham tDCS

SUMMARY:
There are currently no disease-modifying treatments for cognitive and behavioral symptoms associated with early clinical Alzheimer's disease (AD), and only minimally effective symptomatic treatments are available. In this application, we propose a transcranial direct current stimulation (tDCS) augmented executive functioning training intervention. This intervention will target cognition and brain circuits that are impaired in patients with mild cognitive impairment (MCI) and early AD. The goal is to improve cognitive performance and functional outcomes in patients with MCI and early AD.

DETAILED DESCRIPTION:
Objectives There are currently no disease-modifying treatments for cognitive and behavioral symptoms associated with early clinical Alzheimer's disease (AD), and only minimally effective symptomatic treatments are available. In this application, we propose a transcranial direct current stimulation (tDCS) augmented executive functioning training intervention. This intervention will target cognition and brain circuits that are impaired in patients with mild cognitive impairment (MCI) and early AD. The goal is to improve cognitive performance and functional outcomes in patients with MCI and early AD.

Research Plan and Methods This study will recruit 50 Veterans with MCI or very early AD who are receiving outpatient services at the Minneapolis VA Health Care System (MVAHCS) Geriatric Research, Education, and Clinical Center (GRECC) Memory Loss Clinic. This study will be a double-blind, randomized, placebo (sham) controlled study. Participants will be randomly assigned to receive either active or sham tDCS, both paired with cognitive training tasks. Ten sessions of training/tDCS sessions (20 minutes of 2mA current stimulation with 45 minutes of cognitive training tasks) will occur over 2-3 weeks, performed at the participant's home. Participants will attend an in-person enrollment and training session prior to study intervention. Follow-up sessions will occur via phone or video conference at 3 and 6 months after study initiation.

Clinical Relevance Executive cognitive impairments in patients with MCI or early AD have been associated with poor decision-making ability and lack of insight, potentially leading to compromised job performance, financial mismanagement, increased personal safety risk, relationship stress, and poor medical treatment adherence. While disproportionate memory impairment is a hallmark of both conditions, there are compensatory strategies available to reduce disability associated with very early stage memory impairment in those who are otherwise cognitively intact. Compensatory strategies are much less effective for executive dysfunction, as the disability itself impairs one's ability to recognize when such strategies are needed and successfully employ them. Novel, well-tolerated, neuroplasticity-based interventions that can reduce executive impairment by targeting both cognitive control (an executive ability) and its underlying neural dysfunction are needed to improve cognitive outcomes, safety, and quality of life for patients with MCI or early AD. Knowledge gained from this study can inform the future development of clinical treatment approaches aimed at reducing risk and delaying out-of-home placement in Veterans with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study if they:

* are a Veteran receiving services from the MVAHCS GRECC clinic
* have a clinical diagnosis of AD, MCI, or Mild Neurocognitive Disorder presenting as early AD type (predominantly amnestic and dysexecutive)
* are age 60 or older
* are stable on any medications for at least 1 month at the baseline visit
* demonstrate capacity to provide informed consent
* have WiFi access in their home
* have a family member or friend willing to serve as a care partner (care partner needs to have a minimum of 10 hours per week that they see the participant, if they don't live with them).

Exclusion Criteria:

Persons will be excluded from this study if they have:

* any significant medical disorder based on the Principal Investigator's judgment that would impact risk
* other psychiatric or neurological conditions that impact cognition
* metallic cranial plates/screws or implanted devices above the clavicle
* eczema on scalp or other scalp lesions or skin disorders that may become irritated by stimulation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Test of Adult Cognition by Telephone (BTACT) | Change between baseline and 3 week follow-up; 3 and 6 months following study baseline
  Differences in magnitude of change in BTACT scores between active tDCS and sham groups from baseline to follow-up sessions. BTACT covers five cognitive domains: episodic verbal memory (list learning), working memory span (digits backwards), executive functioning (verbal fluency), inductive reasoning (number series completion), and processing speed (backwards counting). Higher total score on the BTACT indicates better cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: John R McCarten, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No